CLINICAL TRIAL: NCT00005338
Title: Homocysteine and Progression of Atherosclerosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4200; R01HL045267 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-12

CONDITIONS: Cardiovascular Diseases; Peripheral Vascular Diseases; Atherosclerosis; Cerebrovascular Disorders; Myocardial Infarction; Heart Diseases; Hyperhomocysteinemia
MeSH Terms: conditions — Cardiovascular Diseases; Peripheral Vascular Diseases; Atherosclerosis; Cerebrovascular Disorders; Myocardial Infarction; Heart Diseases; Hyperhomocysteinemia

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
In the first phase, to establish the relationship of progression of peripheral vascular disease (PVD) to plasma homocysteine. In the second phase, to conduct a randomized, controlled trial of folic acid treatment of plasma homocysteine in peripheral vascular disease.

DETAILED DESCRIPTION:
BACKGROUND:

Few studies of progression of atherosclerotic peripheral vascular disease have been performed and none have used objective methods to evaluate disease progression in a large number of symptomatic subjects. The study is of obvious major clinical importance. Elevated plasma homocysteine is well established as an independent risk factor for atherosclerosis. If folate treatment results in less frequent/rapid progression of peripheral vascular disease, then it will be confirmed as the first effective treatment for atherosclerosis which is without toxic side effects and does not involve major changes in life/dietary habits.

DESIGN NARRATIVE:

The Homocysteine and Progression of Atherosclerosis Study (HPAS) is a long term, prospective, blinded, multifactoral clinical study which began in 1991 to study the relationship between elevated plasma homocysteine (HC) as well as a number of other risk factors and PVD progression. The study is divided into two phases, conducted sequentially upon 400 patients with symptomatic lower extremity (LED) and cerebrovascular disease (CVD). The first phase was a three year natural history study in which relationship of progression of peripheral vascular disease to plasma homocysteine and other risk factors was established. The clinical question addressed by the natural history study was: Do patients with symptomatic peripheral vascular disease and elevated plasma homocysteine have more rapid/frequent progression of peripheral vascular disease than patients with symptomatic peripheral vascular disease and normal plasma homocysteine? Progression of disease was assessed by the primary outcome variables of ankle brachial pressure index and degree of carotid artery stenosis, as determined in the noninvasive vascular laboratory, and by secondary outcome variables including vascular death, need for vascular surgery, stroke, myocardial infarction, amputation, and other clinical events. All outcome variables were determined by investigators blinded to the results of plasma homocysteine testing.

The second phase of the study, which began in August, 1995, is a blinded, prospective, randomized, placebo-controlled trial of folic acid treatment of elevated plasma homocysteine in the same patient population. Folic acid treatment has been demonstrated to result in normalization of elevated plasma homocysteine. The treatment trial addresses the clinical question: Do patients with symptomatic peripheral vascular disease and elevated plasma homocysteine treated with folate have less frequent/rapid progression of peripheral vascular disease than patients with symptomatic peripheral vascular disease and elevated plasma homocysteine treated with placebo? Although the second phase is described as a clinical trial, the Surgery and Bioengineering Study Section describes it as clinical research, not an NIH-defined Phase III trial.

The study was renewed in FY 1999 through 2003 to continue follow-up and analysis.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-08; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lloyd Taylor — Oregon Health and Science University

REFERENCES:
- [Background] McLafferty RB, Moneta GL, Passman MA, Brant BM, Taylor LM Jr, Porter JM. Late clinical and hemodynamic sequelae of isolated calf vein thrombosis. J Vasc Surg. 1998 Jan;27(1):50-6; discussion 56-7. doi: 10.1016/s0741-5214(98)70291-5. PMID 9474082
- [Background] Nehler MR, Taylor LM Jr, Porter JM. Homocysteinemia as a risk factor for atherosclerosis: a review. Cardiovasc Surg. 1997 Dec;5(6):559-67. doi: 10.1016/s0967-2109(97)00062-8. PMID 9423939
- [Background] Abou-Zamzam AM Jr, Lee RW, Moneta GL, Taylor LM Jr, Porter JM. Functional outcome after infrainguinal bypass for limb salvage. J Vasc Surg. 1997 Feb;25(2):287-95; discussion 295-7. doi: 10.1016/s0741-5214(97)70350-1. PMID 9052563
- [Background] Lee RW, Taylor LM Jr, Landry GJ, Goodnight SH, Moneta GL, Edwards JM, Yeager RA, Porter JM. Prospective comparison of infrainguinal bypass grafting in patients with and without antiphospholipid antibodies. J Vasc Surg. 1996 Oct;24(4):524-31; discussion 531-3. doi: 10.1016/s0741-5214(96)70068-x. PMID 8911401
- [Background] McLafferty RB, Moneta GL, Masser PA, Taylor LM Jr, Porter JM. Progression of atherosclerosis in arteries distal to lower extremity revascularizations. J Vasc Surg. 1995 Oct;22(4):450-5; discussion 455-6. doi: 10.1016/s0741-5214(95)70014-5. PMID 7563406
- [Background] McLafferty RB, Moneta GL, Taylor LM Jr, Porter JM. Ability of ankle-brachial index to detect lower-extremity atherosclerotic disease progression. Arch Surg. 1997 Aug;132(8):836-40; discussion 840-1. doi: 10.1001/archsurg.1997.01430320038005. PMID 9267266
- [Background] Deloughery TG, Evans A, Sadeghi A, McWilliams J, Henner WD, Taylor LM Jr, Press RD. Common mutation in methylenetetrahydrofolate reductase. Correlation with homocysteine metabolism and late-onset vascular disease. Circulation. 1996 Dec 15;94(12):3074-8. doi: 10.1161/01.cir.94.12.3074. PMID 8989110
- [Background] Nehler MR, Moneta GL, Lee RW, Edwards JM, Taylor LM Jr, Porter JM. Improving selection of patients with less than 60% asymptomatic internal carotid artery stenosis for follow-up carotid artery duplex scanning. J Vasc Surg. 1996 Oct;24(4):580-5; discussion 585-7. doi: 10.1016/s0741-5214(96)70073-3. PMID 8911406
- [Background] Masser PA, Taylor LM Jr, Porter JM. Importance of elevated plasma homocysteine levels as a risk factor for atherosclerosis. Ann Thorac Surg. 1994 Oct;58(4):1240-6. doi: 10.1016/0003-4975(94)90522-3. PMID 7944799
- [Background] Taylor LM Jr, Chitwood RW, Dalman RL, Sexton G, Goodnight SH, Porter JM. Antiphospholipid antibodies in vascular surgery patients. A cross-sectional study. Ann Surg. 1994 Oct;220(4):544-50; discussion 550-1. doi: 10.1097/00000658-199410000-00012. PMID 7944664
- [Background] Taylor LM Jr, Park TC, Edwards JM, Yeager RA, McConnell DC, Moneta GA, Porter JM. Acute disruption of polytetrafluoroethylene grafts adjacent to axillary anastomoses: a complication of axillofemoral grafting. J Vasc Surg. 1994 Oct;20(4):520-6; discussion 526-8. doi: 10.1016/0741-5214(94)90276-3. PMID 7933253
- [Background] Jacobsen DW, Gatautis VJ, Green R, Robinson K, Savon SR, Secic M, Ji J, Otto JM, Taylor LM Jr. Rapid HPLC determination of total homocysteine and other thiols in serum and plasma: sex differences and correlation with cobalamin and folate concentrations in healthy subjects. Clin Chem. 1994 Jun;40(6):873-81. PMID 8087981
- [Background] Taylor LM Jr, Porter JM. Elevated plasma homocysteine as a risk factor for atherosclerosis. Semin Vasc Surg. 1993 Mar;6(1):36-45. No abstract available. PMID 8252227
- [Background] Nicoloff AD, Taylor LM Jr, McLafferty RB, Moneta GL, Porter JM. Patient recovery after infrainguinal bypass grafting for limb salvage. J Vasc Surg. 1998 Feb;27(2):256-63; discussion 264-6. doi: 10.1016/s0741-5214(98)70356-8. PMID 9510280
- [Background] Taylor LM Jr, Moneta GL, Sexton GJ, Schuff RA, Porter JM. Prospective blinded study of the relationship between plasma homocysteine and progression of symptomatic peripheral arterial disease. J Vasc Surg. 1999 Jan;29(1):8-19; discussion 19-21. doi: 10.1016/s0741-5214(99)70345-9. PMID 9925456
- [Background] Cipolla MJ, Williamson WK, Nehler ML, Taylor LM Jr, Porter JM. The effect of elevated homocysteine levels on adrenergic vasoconstriction of human resistance arteries: the role of the endothelium and reactive oxygen species. J Vasc Surg. 2000 Apr;31(4):751-9. doi: 10.1067/mva.2000.103797. PMID 10753283
- [Background] Lovelace TD, Moneta GL, Abou-Zamzam AM Jr, Edwards JM, Yeager RA, Landry GJ, Taylor LM Jr, Porter JM. Optimizing duplex follow-up in patients with an asymptomatic internal carotid artery stenosis of less than 60%. J Vasc Surg. 2001 Jan;33(1):56-61. doi: 10.1067/mva.2001.112303. PMID 11137924
- [Background] Nicoloff AD, Taylor LM Jr, Sexton GJ, Schuff RA, Edwards JM, Yeager RA, Landry GJ, Moneta GL, Porter JM; Homocysteine and Progression of Atherosclerosis Study Investigators. Relationship between site of initial symptoms and subsequent progression of disease in a prospective study of atherosclerosis progression in patients receiving long-term treatment for symptomatic peripheral arterial disease. J Vasc Surg. 2002 Jan;35(1):38-46; discussion 46-7. PMID 11802131
- [Background] Giswold ME, Landry GJ, Sexton GJ, Yeager RA, Edwards JM, Taylor LM Jr, Moneta GL. Modifiable patient factors are associated with reverse vein graft occlusion in the era of duplex scan surveillance. J Vasc Surg. 2003 Jan;37(1):47-53. doi: 10.1067/mva.2003.4. PMID 12514577
- [Background] Cook JW, Taylor LM, Orloff SL, Landry GJ, Moneta GL, Porter JM. Homocysteine and arterial disease. Experimental mechanisms. Vascul Pharmacol. 2002 May;38(5):293-300. doi: 10.1016/s1537-1891(02)00254-9. PMID 12487034
- [Background] Taylor LM Jr. Elevated plasma homocysteine as risk factor for peripheral arterial disease--what is the evidence? Semin Vasc Surg. 2003 Sep;16(3):215-22. doi: 10.1016/s0895-7967(03)00027-9. PMID 12975761